CLINICAL TRIAL: NCT05523375
Title: Promoting Successful Weight Loss in Primary Care in Louisiana Using Information Technology
Acronym: PROPEL-IT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); University of Alabama at Birmingham (Other); Ochsner Health System (Other)
Responsible Party: Principal Investigator, Peter T. Katzmarzyk, Associate Executive Director for Population and Public Health, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PBRC 2021-072; P50MD017338 (NIH)
Record Dates: First submitted 2022-08-29; First posted 2022-08-31 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Obesity; Diabetes Mellitus, Type 2; PreDiabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Prediabetic State

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intensive Lifestyle Intervention (Experimental): The intervention arm receives a comprehensive, "high-intensity" program, as recommended first-line therapy by the 2013 American Heart Association/American College of Cardiology/The Obesity Society Obesity Guidelines, delivered remotely using eHealth technology, by trained health coaches embedded in the Digital Medicine Group in the Ochsner Health System. The intervention includes remote sessions with the health coach using evidence-based components such as the use of portion control and various behavioral strategies .Patients in the Intervention arm attend weekly sessions in the first six months, followed by monthly sessions for the remaining 18 months.
  Interventions: Behavioral: Intensive Lifestyle Intervention
- Usual Care (No Intervention): Patients in the usual care arm will receive their normal, usual care from their primary care team.

INTERVENTIONS:
Behavioral: Intensive Lifestyle Intervention — Trained health coaches deliver the active intervention - a comprehensive, "high-intensity" program, as recommended first-line therapy by the 2013 American Heart Association/American College of Cardiology/The Obesity Society Guidelines.
  Arms: Intensive Lifestyle Intervention

SUMMARY:
The primary aim is to test the effectiveness of an innovative 24-month pragmatic and scalable weight-loss centric approach using a collaborative care model that connects patients with a non-Primary Care Practitioner (PCP) health coach who delivers care remotely to patients through the patient portal of an electronic medical record (EMR).

DETAILED DESCRIPTION:
This study is a 24-month, two-arm, parallel controlled trial in a primary care setting. A total of 352 Black adults with obesity and type 2 diabetes or prediabetes will be randomized to either 1) intervention or 2) usual care. The intervention arm will receive a comprehensive, "high-intensity" program, as recommended first-line therapy by the 2013 American Heart Association/American College of Cardiology/The Obesity Society Obesity Guidelines, delivered remotely using eHealth technology, by trained health coaches embedded in the Digital Medicine Group in the Ochsner Health System. The intervention will include remote sessions with the health coach using evidence-based components such as the use of portion control and various behavioral strategies. Patients in the usual care arm will receive their normal, usual care from their primary care team. All patients will participate in the collection of patient-reported outcomes at baseline and approximately 6, 12, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* 40-70 years of age
* Self-identify as Black/African American
* Obesity (BMI 30.0-50.0 kg/m2)
* Type II diabetes (based on ICD-10 codes, fasting plasma glucose ≥126 mg/dL, HbA1c ≥6.5%, 2-h plasma glucose during 75-g Oral Glucose Tolerance Test (OGTT) ≥200 mg/dL, or a random plasma glucose ≥200 mg/dL in a patient with classic symptoms of hyperglycemia or hyperglycemic crisis) or pre-diabetes (based on ICD-10 codes, fasting glucose 100-125 mg/dL or HbA1c 5.7-6.4% or 2-h glucose during 75-g OGTT 140-199 mg/dL)
* Has an internet-connected device and is willing to use it for intervention delivery
* Patient in the Ochsner Health System with an active MyOchsner portal account, or willing to create one
* Acknowledgement from their Ochsner primary care practitioner that there are no known contraindications to the patient's participation
* Have weight measured at an Ochsner clinic within 4 weeks of screening
* Resident of Louisiana
* Be able to provide informed consent
* Willing to change diet and/or physical activity

Exclusion Criteria:

* Body weight ≥ 400 lbs.
* Current use of weight loss medication or recent weight loss (net loss >10 lbs in the last six months)
* Currently participating in a structured weight loss program
* Plans to move from the area within 2 years
* Given birth within the past year, is currently pregnant or breastfeeding or plans to become pregnant within 2 years
* Past bariatric surgery or plans for bariatric surgery within 2 years
* Disease/condition that is life threatening or can interfere with or be aggravated by exercise or weight loss

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2022-08-29 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Body weight (Percent Change) | Percent (%) Change from Baseline to Month 24
  Body weight is measured in light indoor clothes and is obtained from the electronic medical record.

SECONDARY OUTCOMES:
Body weight (kg) | Change in kg from Baseline to Month 24
  Body weight is measured in light indoor clothes and is obtained from the electronic medical record.
Systolic Blood Pressure | Change from Baseline to Month 24
  Resting systolic blood pressure is measured and is obtained from the electronic medical record.
Diastolic Blood Pressure | Change from Baseline to Month 24
  Resting diastolic blood pressure is measured and is obtained from the electronic medical record.
HbA1c | Change from Baseline to Month 24
  HbA1c levels are assayed and are obtained from the electronic medical record.
Total Cholesterol | Change from Baseline to Month 24
  Total cholesterol levels are assayed and are obtained from the electronic medical record.
High-density Lipoprotein (HDL) Cholesterol | Change from Baseline to Month 24
  HDL cholesterol levels are assayed and are obtained from the electronic medical record.
Triglycerides | Change from Baseline to Month 24
  Triglyceride levels are assayed and are obtained from the electronic medical record.
Low-density Lipoprotein (LDL) cholesterol | Change from Baseline to Month 24
  LDL cholesterol levels are estimated using the Friedewald equation and are obtained from the electronic medical record.
Physical Activity | Change from Baseline to Month 24
  Physical activity is measured using the International Physical Activity Questionnaire-SF questionnaire.
Dietary Intake | Change from Baseline to Month 24
  Dietary intake is measured using National Cancer Institute Dietary Screeners.
Impact of Weight on Quality of Life-Lite-Clinical Trials Questionnaire | Change from Baseline to Month 24
  Items are scored 1-5 (never true to completely true). Scores are obtained on 3 composite scales (Physical, Physical Function, and Psychosocial), as well as total score. The raw composite score is calculated as the average of non-missing responses within each composite, then transforming to a 0-100 scale (worst to best). Composite scores and total score range from 0 to 100, where 100 represents higher levels of functioning.
EuroQol-5 Dimension Questionnaire | Change from Baseline to Month 24
  Each of 5 questions can have a response ranging from 1-5 (none to extreme). These are then concatenated into one of 3125 "health states" (i.e. 11231, 52454, etc.) An EQ-5D summary index is derived by applying a formula that attaches values (weights) to each of the levels in each dimension to create a value set. Lower scores indicate better health.
Health Care Utilization Questionnaire | Change from Baseline to Month 24
  Health care utilization is measured using a brief 4-item questionnaire with continuous responses (how many times did you go to the doctor, go to Emergency Room, stay overnight, # nights). Each question is analyzed separately.
Perceived Stress Scale-4 Questionnaire | Change from Baseline to Month 24
  The Perceived Stress Scale has 4 questions with responses ranging from 0-4 (Never to Very Often). Total (sum) score range is 0-16, with a higher score correlating to more stress.

CONTACTS AND LOCATIONS:
Overall Officials: Peter T Katzmarzyk, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified individual-level dataset will be made available to researchers making a reasonable request and upon approval of the PROPEL-IT Publications Committee. Data will be made available 1 year after publication of the primary outcomes manuscript.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available upon reasonable request to the Principal Investigator 1 year after the publication of the Primary Outcomes manuscript for up to 5 years.
Access Criteria: Access to the data must be approved by the PROPEL-IT Publications Committee.

REFERENCES:
- [Derived] Katzmarzyk PT, Price-Haywood EG, Apolzan JW, Denstel KD, Drews KL, Farris E, Harden-Barrios J, Hearld LR, Mire EF, Martin CK, Newton RL, Pisu M. Improving weight loss and cardiometabolic risk in black patients with diabetes or pre-diabetes: Rationale and protocol for a digital medicine hybrid type 1 implementation trial. Contemp Clin Trials. 2025 Feb;149:107806. doi: 10.1016/j.cct.2024.107806. Epub 2025 Jan 3. PMID 39756673